CLINICAL TRIAL: NCT06806501
Title: Muscle Mass, Quality, and the Menopause: Sex-specific Strategies to Mitigate Sarcopenia in Ageing Populations
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Matthew Brook, Associate Professor, University of Nottingham
Other Study IDs: FMHS 129-0224
Record Dates: First submitted 2024-06-18; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premenopausal: Defined as having a menstrual cycle and having plasma follicle-stimulating hormone (FSH) <30 IU/L, taken during days 1-5 of their menstrual cycle.
  Interventions: Behavioral: Unilateral Resistance Exercise
- Postmenopausal: Defined as having no menses for 12 months, E2 (Oestradiol) < 118pmol/L and FSH >30 IU/L.
  Interventions: Behavioral: Unilateral Resistance Exercise

INTERVENTIONS:
Behavioral: Unilateral Resistance Exercise — Resistance exercise training session, consisting of 6 x 8 repetitions of leg extension (of the non-dominant leg) at 75% 1RM (repetition maximum) with 2 min rest between sets.

SUMMARY:
Aging causes muscles to often become smaller and weaker resulting in physical frailty and functional impairments, such as difficulty raising from a chair, dressing, and preparing meals. In the UK there is a growing aged population with those >65y expected to increase from 18% of the population in 2016, to 26% by 2066. As such, age related muscle mass loss and functional impairments represents one of the largest problems facing the health care services. There is an urgent need to develop strategies to reduce healthcare costs and improve health and wellbeing with age. These strategies must be targeted, as evidence suggests that the loss in muscle size and strength is different between men and women throughout the aging process. For example, older women have greater levels of physical disability that includes difficulties in walking around the home, getting out of a bed or chair, and eating, compared with men. These sex differences with ageing are unclear, yet the greater levels of physical disability could be the result of the menopause. The menopause describes a change in the sex hormone environment that is a part of normal female ageing. Physical disability can be further enhanced by an increase in body fat during the menopause in the face of decreasing muscle mass. Currently, there is a lack of understanding as to how these changes in body composition occur, with no effective treatments against muscle mass loss. The aims of this project are to increase understanding on how the menopause impacts muscle mass regulation. In addition, the investigators will use novel magnetic resonance imaging (MRI) techniques to map the distribution of newly created fat, and qualitative interviews to better understand how resistance exercise therapy (RET) can be incorporated into the daily lives of postmenopausal women.

DETAILED DESCRIPTION:
The age-related loss of muscle mass and function (sarcopenia) inevitably results in physical frailty and functional impairments, such as difficulty raising from a chair, dressing, and preparing meals. With a rapidly growing aged population (those >65y increasing from 18% of the population in 2016, to 26% by 2066), sarcopenia represents one of the largest problems facing health care services. Excess healthcare costs associated with sarcopenia are rapidly growing and were estimated to be £2.5 billion in 2016. There is an urgent need to develop strategies to mitigate sarcopenia to reduce healthcare costs and improve health and wellbeing with age. These strategies must be targeted, as evidence suggests that there is sexual dimorphism in ageing and the development of sarcopenia. Sarcopenia develops earlier in women, resulting in greater levels of physical disability that includes difficulties in walking, getting out of a chair, and eating, compared with men. The mechanistic sex differences with ageing are unclear, yet the earlier prevalence of sarcopenia in women coincides with the menopause. In addition, physical disability can be further exacerbated by an increase in adiposity during the menopause in the face of decreasing muscle mass. This change in body composition includes ectopic fat infiltration into muscle that is associated with decreased muscle performance, however, currently, there is a lack of understanding as to how these changes in body composition occur.

Understanding the underlying mechanisms that bring about change in physiological systems is key in the development of interventions. Muscle mass is controlled by the balance between muscle protein synthesis (MPS) and muscle protein breakdown (MPB). With age, many of the signals that increase MPS (i.e., nutrient intake and activity) become less effective, resulting in negative protein balance and muscle loss. Since muscle loss is accelerated after the menopause in women, there must be a greater imbalance between MPS and MPB. The measurement of MPS and MPB can be achieved using stable isotope tracer techniques that can be followed throughout the body. However, there is a lack of research into the mechanistic effects of the menopause on muscle mass regulation. In addition to measures of muscle protein turnover, the investigators have recently used stable isotope tracer techniques alongside MRI scanning to image deuterium incorporation within lipid. the investigators will use these techniques to image newly created fat to further understanding of body composition changes in post-menopausal women.

Resistance exercise therapy (RET) currently offers the most effective strategy to mitigate muscle mass loss and improve body composition with ageing, by increasing MPS, promoting muscle hypertrophy, and building strength8. However, older women display blunted muscle hypertrophy in response to RET (when compared to younger women, and older men), and it is not known how the menopause affects hypertrophic responses to exercise. Further, for any intervention to have a meaningful impact, it must be effectively incorporated by postmenopausal women into their daily lives. The investigators have conducted an evaluation of physical activity interventions for post-menopausal women, which revealed that women going through the menopause want more evidence-based guidance on how much and what type of exercise they should be doing, and on whether exercise can alleviate menopausal symptoms and prevent muscle loss.

Aims: To investigate the effects of the menopause on muscle mass regulation, changes in body composition, and assess the acceptability and effectiveness of RET.

ELIGIBILITY:
Inclusion Criteria:

* Biological woman, 18-65 years of age
* Body mass index (BMI) 18-30 kg/m2
* Non smoker
* Not performing regular resistance type exercise
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* A BMI <18 or >39 kg·m-2
* Active cardiovascular disease: uncontrolled hypertension (Blood pressure > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt or recent cardiac event.
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial)
* Respiratory disease including pulmonary hypertension or Chronic obstructive pulmonary disease (COPD).
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes (treated and untreated), polycystic ovarian syndrome (PCOS), inborn/ congenital errors of metabolism (e.g. Phenylketonuria (PKU), galactosaemia)
* Active inflammatory bowel disease.
* Acute infection.
* Acute or chronic renal disease.
* Malignancy (or history of malignancy with 5 y).
* Recent (within 6 mo) or current steroid treatment, hormone replacement therapy (HRT), hormonal contraception, or other hormonal therapies that may interfere with outcome measures.
* Coagulopathy.
* Musculoskeletal or neurological disorders.
* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.
* Amenorrhoea for a reason other than menopause.
* Contraindications for Magnetic Resonance Imaging (MRI).
* Allergy or sensitivity to local anaesthesia, or dressing adhesive.
* Inner ear pathology or vertigo

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be healthy females aged 18 - 65, who are not on hormonal replacement therapy or hormonal contraceptives and are not participating in regular resistance exercise.
  Participants will fall into two groups:
  * Premenopausal, defined as having a menstrual cycle and having plasma follicle-stimulating hormone (FSH) <30 IU/L, taken during days 1-5 of their menstrual cycle.
  * Postmenopausal, defined as having no menses for 12 months, E2 (Oestradiol) < 118pmol/L and FSH >30 IU/L.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of muscle protein synthesis | 3 Days
  Comparison between pre and post menopausal women of vastus lateralis muscle protein synthesis in response to acute unilateral resistance exercise and at rest using deuterium oxide stable isotope techniques.
Rate of muscle protein breakdown | 3 Days
  Comparison between pre and post menopausal women of whole body muscle protein breakdown in response to acute unilateral resistance exercise and at rest using D3-3-methylhistidine

SECONDARY OUTCOMES:
Whole body muscle mass | At the point of enrolment
  Comparison between pre and post menopausal women of whole body muscle mass using D3-Creatine
Quadriceps fat mass | At the point of enrolment
  Comparison between pre and post menopausal women of quadriceps fat using Dixon magnetic resonance imaging (MRI) of the quadriceps
Menopausal symptoms | At the point of enrolment
  Comparison between pre and post menopausal women of menopausal symptoms on the menopause rating scale (0 - 44; higher score = greater menopause symptoms)
Knee extensor strength | At the point of enrolment
  Comparison between pre and post menopausal women of knee extensor muscle strength in response to unilateral exercise training using a cybex dynamometer
De novo lipogenesis | 0 - 8 weeks
  Use deuterium magnetic resonance imaging (MRI) to map the distribution of newly created lipid in pre and post menopausal women.
Intramuscular protein signalling | 0 - 3 Days
  Comparison between pre and post menopausal women of intramuscular protein signalling in response to unilateral resistance exercise using immunoblotting.
Muscle gene expression | 0 - 3 Days
  Comparison between pre and post menopausal women of muscle messenger ribonucleic acid (mRNA) gene expression in response to unilateral resistance exercise using polymerase chain reactions (PCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Queens Medical Centre Campus, Nottingham, United Kingdom